CLINICAL TRIAL: NCT01802385
Title: Adjunctive Sertraline for the Treatment of HIV-Associated Cryptococcal Meningitis
Acronym: ASTRO-CM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Infectious Disease Institute, Kampala, Uganda (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Mbarara University of Science and Technology (Other); Medical Research Council (Other Government); Wellcome Trust (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S4 0296-01; R01NS086312-01 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cryptococcal Meningitis; Fungal Meningitis
Keywords: cryptococcal meningitis; cryptococcus; meningitis; yeast; fungus
MeSH Terms: conditions — Meningitis, Cryptococcal; Meningitis, Fungal; Meningitis | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (No Intervention): Standard cryptococcal meningitis therapy with amphotericin (0.7-1.0 mg/kg/day) + fluconazole (800-1200mg/day) + placebo
- Sertraline 400mg (Experimental): Standard cryptococcal meningitis therapy with amphotericin (0.7-1.0 mg/kg/day) + fluconazole (800-1200mg/day plus adjunctive sertraline therapy at 400mg/day for 2 weeks, then 200mg for 12 weeks, and then tapered over 3 weeks.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Sertraline 400mg/day for 2 weeks, then 200mg/day for 12 weeks, then tapered over 3 weeks.
  Other Names: Zoloft; Lustral
  Arms: Sertraline 400mg

SUMMARY:
This is a phase III trial to determine whether adjunctive sertraline will lead to improved survival 18-week survival.

There was an initial phase I/II unmasked dose finding pharmacokinetic study of CSF concentrations in 172 persons conducted from August 2013 to August 2014. See NCT03002012.

DETAILED DESCRIPTION:
This is a phase III randomized trial to evaluate whether sertraline when added to standard amphotericin-based therapy for cryptococcal meningitis, will lead to improved survival . Cryptococcal meningitis diagnosis will be made via CSF cryptococcal antigen (CRAG) at time of lumbar puncture (LP) with confirmation by CSF culture. After informed consent, subjects that meet eligibility requirements will be able to enter study. A non-randomized phase I dose-escalation study will first be conducted to help optimize dosing for a larger randomized phase II study.

Phase III Design: Subjects will be randomized to standard induction therapy with masked placebo or sertraline at 400mg/day. We will use a permutated block randomization in a 1:1 allocation (n=275 per arm). Total anticipated enrollment: 550 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Cryptococcal meningitis diagnosed by CSF cryptococcal antigen (CRAG)
* HIV-1 infection
* Ability and willingness of the participant or legal guardian/representative to provide informed consent
* Willing to receive protocol-specified lumbar punctures

Exclusion Criteria:

* Age < 18 years
* Receipt of >=3 doses of amphotericin therapy
* Cannot or unlikely to attend regular clinic visits
* History of known liver cirrhosis
* Presence of jaundice
* Pregnancy
* Current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Meya, MBCHB MMed, Principal Investigator — Infectious Disease Institute; Joshua Rhein, MD, Study Director — University of Minnesota; David R Boulware, MD MPH, Study Chair — University of Minnesota
Locations (2):
- Uganda (2):
  - Infectious Disease Institute, Kampala
  - Mbarara University of Science and Technology, Mbarara

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Open
Access Criteria: Contact of the Principal Investigator

REFERENCES:
- [Background] Rhein J, Morawski BM, Hullsiek KH, Nabeta HW, Kiggundu R, Tugume L, Musubire A, Akampurira A, Smith KD, Alhadab A, Williams DA, Abassi M, Bahr NC, Velamakanni SS, Fisher J, Nielsen K, Meya DB, Boulware DR; ASTRO-CM Study Team. Efficacy of adjunctive sertraline for the treatment of HIV-associated cryptococcal meningitis: an open-label dose-ranging study. Lancet Infect Dis. 2016 Jul;16(7):809-818. doi: 10.1016/S1473-3099(16)00074-8. Epub 2016 Mar 10. PMID 26971081
- [Background] Zhai B, Wu C, Wang L, Sachs MS, Lin X. The antidepressant sertraline provides a promising therapeutic option for neurotropic cryptococcal infections. Antimicrob Agents Chemother. 2012 Jul;56(7):3758-66. doi: 10.1128/AAC.00212-12. Epub 2012 Apr 16. PMID 22508310
- [Background] Smith KD, Achan B, Hullsiek KH, McDonald TR, Okagaki LH, Alhadab AA, Akampurira A, Rhein JR, Meya DB, Boulware DR, Nielsen K; ASTRO-CM/COAT Team. Increased Antifungal Drug Resistance in Clinical Isolates of Cryptococcus neoformans in Uganda. Antimicrob Agents Chemother. 2015 Dec;59(12):7197-204. doi: 10.1128/AAC.01299-15. Epub 2015 Aug 31. PMID 26324276
- [Result] Rhein J, Huppler Hullsiek K, Tugume L, Nuwagira E, Mpoza E, Evans EE, Kiggundu R, Pastick KA, Ssebambulidde K, Akampurira A, Williams DA, Bangdiwala AS, Abassi M, Musubire AK, Nicol MR, Muzoora C, Meya DB, Boulware DR; ASTRO-CM team. Adjunctive sertraline for HIV-associated cryptococcal meningitis: a randomised, placebo-controlled, double-blind phase 3 trial. Lancet Infect Dis. 2019 Aug;19(8):843-851. doi: 10.1016/S1473-3099(19)30127-6. PMID 31345462
- [Derived] Sadiq A, Kwizera R, Kiiza TK, Ayebare P, Ahimbisibwe C, Ndyetukira JF, Boulware DR, Meya DB. Experiences, challenges, gaps, and strategies for counselling persons presenting with advanced HIV-associated meningitis in Uganda. AIDS Res Ther. 2025 Feb 19;22(1):21. doi: 10.1186/s12981-025-00705-z. PMID 39972326
- [Derived] Okurut S, Boulware DR, Okafor E, Rhein J, Kajumbula H, Bagaya BS, Bwanga F, Olobo JO, Manabe YC, Meya DB, Janoff EN. Divergent neuroimmune signatures in the cerebrospinal fluid predict differential gender-specific survival among patients with HIV-associated cryptococcal meningitis. Front Immunol. 2023 Dec 13;14:1275443. doi: 10.3389/fimmu.2023.1275443. eCollection 2023. PMID 38152404
- [Derived] Bahr NC, Skipper CP, Huppler-Hullsiek K, Ssebambulidde K, Morawski BM, Engen NW, Nuwagira E, Quinn CM, Ramachandran PS, Evans EE, Lofgren SM, Abassi M, Muzoora C, Wilson MR, Meya DB, Rhein J, Boulware DR. Recurrence of Symptoms Following Cryptococcal Meningitis: Characterizing a Diagnostic Conundrum With Multiple Etiologies. Clin Infect Dis. 2023 Mar 21;76(6):1080-1087. doi: 10.1093/cid/ciac853. PMID 36303432
- [Derived] Lofgren SM, Nicol MR, Kandole TK, Castillo-Mancilla J, Anderson PL, Mpoza E, Tugume L, Bangdiwala AS, Ssebambulidde K, Hullsiek KH, Rhein J, Meya DB, Boulware DR. Short Communication: A Descriptive Analysis of Dried Blood Spot Adherence Testing Among Ugandans with HIV Presenting with Cryptococcal Meningitis. AIDS Res Hum Retroviruses. 2021 Jul;37(7):529-533. doi: 10.1089/AID.2020.0202. Epub 2021 Apr 12. PMID 33677986
- [Derived] Kwizera R, Sadiq A, Ndyetukira JF, Nalintya E, Williams D, Rhein J, Boulware DR, Meya DB; COAT and ASTRO trial teams. Impact of community engagement and social support on the outcomes of HIV-related meningitis clinical trials in a resource-limited setting. Res Involv Engagem. 2020 Aug 20;6:49. doi: 10.1186/s40900-020-00228-z. eCollection 2020. PMID 32843994
- [Derived] Ahimbisibwe C, Kwizera R, Ndyetukira JF, Kugonza F, Sadiq A, Hullsiek KH, Williams DA, Rhein J, Boulware DR, Meya DB. Management of amphotericin-induced phlebitis among HIV patients with cryptococcal meningitis in a resource-limited setting: a prospective cohort study. BMC Infect Dis. 2019 Jun 26;19(1):558. doi: 10.1186/s12879-019-4209-7. PMID 31242860
- [Derived] Atherton RR, Ellis J, Cresswell FV, Rhein J, Boulware DR. Ophthalmic signs in Ugandan adults with HIV-associated cryptococcal meningitis: A nested analysis of the ASTRO-CM cohort. Wellcome Open Res. 2018 Oct 12;3:80. doi: 10.12688/wellcomeopenres.14666.2. eCollection 2018. PMID 30345376
- [Derived] Tugume L, Rhein J, Hullsiek KH, Mpoza E, Kiggundu R, Ssebambulidde K, Schutz C, Taseera K, Williams DA, Abassi M, Muzoora C, Musubire AK, Meintjes G, Meya DB, Boulware DR; COAT and ASTRO-CM teams. HIV-Associated Cryptococcal Meningitis Occurring at Relatively Higher CD4 Counts. J Infect Dis. 2019 Feb 23;219(6):877-883. doi: 10.1093/infdis/jiy602. PMID 30325463
- [Derived] Ssebambulidde K, Bangdiwala AS, Kwizera R, Kandole TK, Tugume L, Kiggundu R, Mpoza E, Nuwagira E, Williams DA, Lofgren SM, Abassi M, Musubire AK, Cresswell FV, Rhein J, Muzoora C, Hullsiek KH, Boulware DR, Meya DB; Adjunctive Sertraline for Treatment of HIV-associated Cryptococcal Meningitis Team. Symptomatic Cryptococcal Antigenemia Presenting as Early Cryptococcal Meningitis With Negative Cerebral Spinal Fluid Analysis. Clin Infect Dis. 2019 May 30;68(12):2094-2098. doi: 10.1093/cid/ciy817. PMID 30256903
- See also: Infectious Disease Institute — http://www.idi-makerere.com/
- See also: Accordia Global Health Foundation — http://www.accordiafoundation.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Standard cryptococcal meningitis therapy with amphotericin (0.7-1.0 mg/kg/day) + fluconazole (800-1200mg/day).
  Sertraline: Sertraline 400mg/day for 2 weeks, then 200mg/day for 12 weeks, then tapered over 3 weeks.
Period: Overall Study
Arm/Group | Placebo | Sertraline 400mg
Started | 231 | 229
Completed | 125 | 109
Not Completed | 106 | 120
Not completed — Death | 106 | 120

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sertraline 400mg | Total
Number analyzed (Participants) | 231 | 229 | 460
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 231 | 229 | 460
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [30 to 41] | 35 [29 to 40] | 35 [30 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 97 | 184
  Male | 144 | 132 | 276
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 231 | 229 | 460
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 231 | 229 | 460

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: 18-week survival. The comparison will be between sertraline 400mg group and placebo
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
Participants | 125 | 109

2. Secondary Outcome: Safety (Occurence of Adverse Events)
Description: Safety and tolerability of adjunctive sertraline (grade 4-5) adverse reactions
Time Frame: 18 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
events | 121 | 141

3. Secondary Outcome: Count of Participants With Cerebrospinal Fluid Sterility
Description: Number of participants with sterile cerebrospinal fluid at 2 weeks
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
Participants | 90 | 101

4. Secondary Outcome: Center for Epidemiologic Studies in Depression (CES-D) Scale
Description: Center for Epidemiologic Studies in Depression (CES-D) scale at 14 weeks. CES-D scores are based on a 20 item survey with total scores ranging from 0 to 60. Higher scores suggest a greater presence of depressive symptoms. A CES-D score of 16 or higher is interpreted to indicate a risk for depression.
Time Frame: 14 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
score on a scale | 16.6 [14.3 to 18.8] | 13.2 [11.0 to 15.5]

5. Secondary Outcome: Quantitative Neurocognitive Performance Score (QNPZ-8)
Description: Quantitative neurocognitive performance Z-score (QNPZ-8) at 14 weeks. The QNPZ-8 is a mean score of testing of 8 neurocognitive domains. Eqach domain is scaled based on a Z-score where the mean = 0 for the HIV-negative Ugandan population, accounting for age and educational status. Each +1 unit is one standard deviation better than the population norm. Each -1 unit is one standard deviation worse than the population norm.
Time Frame: 14 weeks
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
score | -1.4 [-1.5 to -1.2] | -1.3 [-1.4 to 1.1]

6. Secondary Outcome: Fungal Clearance as Determined by Early Fungicidal Activity of CDF
Description: To determine whether adjunctive sertraline will lead to a faster rate of fungal clearance from cerebrospinal fluid (CSF), as measured by early fungicidal activity (EFA) of clearance of the Cryptococcus colony forming units (cfu) per mL of CSF per day, compared to standard therapy alone.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: -log10 CFU/ml/day
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
-log10 CFU/ml/day
  General Linear Regression | 0.47 [0.4 to 0.54] | .43 [.37 to .50]
  Mixed-Effects Regression | 0.33 [.3 to .35] | .33 [.3 to .36]

7. Secondary Outcome: Number of Participants Experiencing IRIS OR Relapse
Description: Cumulative incidence of central nervous system (CNS) cryptococcal-related paradoxical immune reconstitution inflammatory syndrome (IRIS) or culture-positive relapse
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
Participants | 9 | 5

8. Secondary Outcome: Event Free Survival
Description: Event free survival of composite events of: death,central nervous system (CNS) cryptococcal-related paradoxical immune reconstitution inflammatory syndrome (IRIS) or culture-positive relapse.
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sertraline 400mg
Number analyzed (Participants) | 231 | 229
Participants | 116 | 103

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Serious adverse events were collected on a condition-by-condition basis. Non-serious adverse event information was assessed in such a manner that the specific Adverse Event Terms cannot be separated.
Arm/Group | Placebo | Sertraline 400mg
All-Cause Mortality (participants affected / at risk) | 106/231 | 120/229
Serious Adverse Events (participants affected / at risk) | 121/231 | 141/229
Other Adverse Events (participants affected / at risk) | 65/231 | 66/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=231) | Sertraline 400mg (N=229)
Fever (General disorders) | 4 | 1
Infection (Infections and infestations) | 3 | 1
Hypotension (General disorders) | 1 | 2
Thrombosis (Blood and lymphatic system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Altered Mental Status (Psychiatric disorders) | 1 | 3
Headache (General disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Elevated Creatinine (Blood and lymphatic system disorders) | 9 | 13
Hypokalemia (Blood and lymphatic system disorders) | 4 | 13
Hyperkalemia (Blood and lymphatic system disorders) | 2 | 0
Hyponatremia (Blood and lymphatic system disorders) | 13 | 16
Hypernatremia (Blood and lymphatic system disorders) | 0 | 2
Hypomagnesemia (Blood and lymphatic system disorders) | 2 | 0
Acidosis (Blood and lymphatic system disorders) | 0 | 3
Anemia (Blood and lymphatic system disorders) | 49 | 54
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 9 | 10
Elevated ALT (Blood and lymphatic system disorders) | 2 | 0
Elevated AST (Blood and lymphatic system disorders) | 3 | 0
Elevated Bilirubin (Blood and lymphatic system disorders) | 10 | 9
Anorexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=231) | Sertraline 400mg (N=229)
Non-serious Adverse Events (General disorders) | 65 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT01802385/Prot_SAP_000.pdf